CLINICAL TRIAL: NCT05567055
Title: A Phase 2 Open-label Study to Determine the Central Nervous System Efficacy of Capmatinib in NSCLC Patients With Brain Metastases With cfDNA Positive MET Alterations
Brief Title: Central Nervous System Efficacy of Capmatinib in NSCLC With Brain Metastases With cfDNA Positive MET Alterations
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Timothy Burns, MD, PHD (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor-Investigator, Timothy Burns, MD, PHD, Associate Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCC 22-010
Record Dates: First submitted 2022-09-30; First posted 2022-10-05 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Non-small Cell Lung Cancer
Keywords: cfDNA positive MET alterations; MET amplification; METΔex14 mutation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — capmatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Capmatinib (Experimental): 400 mg orally, twice daily
  Interventions: Drug: Capmatinib

INTERVENTIONS:
Drug: Capmatinib — Capmatinib is a medication for the treatment of metastatic non-small cell lung cancer tumors that have a mutation that leads to the exon 14 skipping of the MET gene, which codes for the membrane receptor HGFR
  Other Names: Tabrecta

SUMMARY:
This is a phase II single-arm open label trial to evaluate the intracranial efficacy of capmatinib in advanced stage NSCLC with asymptomatic BM with positive MET amplification or METΔex14 detected on cfDNA.

DETAILED DESCRIPTION:
This will be a phase II single-arm open label trial of capmatinib at a dose of 400 mg orally twice daily in advanced stage NSCLC with asymptomatic BM with positive MET amplification or METΔex14 detected on cfDNA. This trial will evaluate the intracranial efficacy of capmatinib in cfDNA MET amplification or mutation positive NSCLC. Potentially eligible patients will undergo prescreening with Predicine's cfDNA assay to identify cfDNA MET amplification or mutation positive NSCLC patients. Radiographic assessments for cranial and extracranial disease response will occur every 8 weeks. Capmatinib will be given until disease progression or intolerability of treatment. A two-stage single arm design will be used to establish whether the proportion of responses is sufficiently high to warrant further testing and to allow stopping for futility at the first stage.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. Written informed consent and any locally required authorization (e.g., Health Insurance Portability and Accountability Act in the US, European Union [EU] Data Privacy Directive in the EU) obtained from the patient/legal representative prior to performing any protocol-related procedures, including screening evaluations.
2. Age >18 years at time of study entry.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. Adequate normal organ and marrow function as defined below:

   1. Absolute neutrophil count (ANC) ≥ 1.5 x 109/L without growth factor support
   2. Platelets ≥ 100 x 109/L
   3. Hemoglobin (Hgb) ≥ 9 g/dL
   4. Calculated creatinine clearance (using Cockcroft-Gault formula) ≥ 45 mL/min
   5. Total bilirubin (TBIL) ≤ 1.5 x ULN (upper limit of normal)
   6. Aspartate transaminase (AST) ≤ 3 x ULN, except for patients with liver metastasis, who may only be included if AST ≤ 5 x ULN
   7. Alanine transaminase (ALT) ≤ 3 x ULN, except for patients with liver metastasis, who may only be included if ALT ≤ 5 x ULN
   8. Alkaline phosphatase (ALP) ≤ 5.0 x UL
   9. Asymptomatic serum amylase ≤ Grade 2. Patients with Grade 1 or Grade 2 serum amylase at the beginning of the study must be confirmed to have no signs and/or symptoms suggesting pancreatitis or pancreatic injury (e.g. elevated P-amylase, abnormal imaging findings of pancreas, etc.)
   10. Serum lipase ≤ ULN
5. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
6. Participants must have a life expectancy of at least 3 months
7. Confirmed histologic or cytologic diagnosis of Stage IV non-squamous NSCLC.
8. Untreated asymptomatic brain metastases must be > 1 measurable CNS lesion per RANO-BM (> 10mm) which is asymptomatic in the absence of steroids. Prior radiation is allowed if progression has been documented after radiation and only radiation necrosis or pseudoprogression is unlikely.
9. Capable of undergoing magnetic resonance imaging (MRI).
10. Positive for MET amplification or METΔex14 mutation using Predicine's cfDNA assay (PredicineCARE). Patients with detection of MET amplification or METΔex14 mutation utilizing an alternative CLIA certified blood based ctDNA or cfDNA assay may be allowed at the discretion of the PI.
11. Available archival tissue or able to undergo a biopsy.
12. Any number of lines of prior therapy are allowable.

Exclusion Criteria:

1. Treatment with prior MET tyrosine kinase inhibitor or HGF-targeting therapy. Treatment with other MET targeted therapies such as monoclonal antibodies may be allowed at the discretion of the PI.
2. Prior SRS or WBXRT without evidence of CNS progression.
3. Participants who are receiving concomitant corticosteroids must be on a stable or decreasing dose for at least 1 month prior to the first dose of study treatment. If patients are on corticosteroids for endocrine deficiencies or tumor-associated symptoms other than CNS related, dose must have been stabilized (or decreasing) for at least 5 days before first dose of capmatinib. Note: dose of steroids must be stable for 5 days before the baseline brain MRI.
4. Patient with symptomatic brain metastases or leptomeningeal disease are excluded. Patients with asymptomatic leptomeningeal disease may be allowed at the principal investigator's discretion.
5. Presence or history of a malignant disease other than NSCLC that has been diagnosed and required therapy within the past 3 years. Exceptions to this exclusion include: completely resected basal cell and squamous cell skin cancers, and completely resected carcinoma in situ of any type.
6. Participants with other known targetable molecular alterations (such as ROS1, RET, NTRK1-3 translocations or BRAF mutation) who might be candidates to alternative targeted therapies as applicable per local regulations and treatment guidelines
7. Participants with EGFR mutant and ALK fusion positive NSCLC are excluded.
8. Presence or history of interstitial lung disease or interstitial pneumonitis, including clinically significant radiation pneumonitis (i.e., affecting activities of daily living or requiring therapeutic intervention)
9. Clinically significant, uncontrolled heart diseases including:

   1. Unstable angina within 6 months prior to screening
   2. Myocardial infarction within 6 months prior to screening
   3. History of documented congestive heart failure (New York Heart Association functional classification III-IV)
   4. Uncontrolled hypertension defined by a Systolic Blood Pressure (SBP) ≥ 160 mm Hg and/or Diastolic Blood Pressure (DBP) ≥ 100 mm Hg, with or without antihypertensive medication. Initiation or adjustment of antihypertensive medication(s) is allowed prior to enrolment
   5. Ventricular arrhythmias
   6. Supraventricular and nodal arrhythmias not controlled with medication
   7. Other cardiac arrhythmia not controlled with medication
   8. QTcF ≥ 470 ms on the screening ECG (as mean of triplicate ECG)
   9. History of familial long QT syndrome, sudden death or congenital long QT syndrome
10. Thoracic radiotherapy to lung fields ≤ 4 weeks prior to starting capmatinib or subjects who have not recovered from radiotherapy-related toxicities. For all other anatomic sites (including radiotherapy to thoracic vertebrae and ribs), radiotherapy ≤ 2 weeks prior to starting capmatinib or subjects who have not recovered from clinically significant radiotherapy-related toxicities. Palliative radiotherapy for bone lesions ≤ 2 weeks prior to starting capmatinib is allowed.
11. Major surgery (e.g., intra-thoracic, intra-abdominal or intra-pelvic) within 4 weeks prior to starting study treatment (2 weeks for resection of brain metastases) or subjects who have not recovered from the side effects of such a procedure. Video-assisted thoracic surgery (VATS) and mediastinoscopy will not be counted as major surgery and subjects can be enrolled in the study ≥1 week after the procedure
12. Participants receiving treatment with strong inducers of CYP3A and could not be discontinued at least 1 week prior to the start of treatment with capmatinib and for the duration of the study.
13. Participants receiving treatment with any enzyme-inducing anticonvulsant that cannot be discontinued at least 1 week before first dose of capmatinib, and for the duration of the study. Participants on non-enzyme-inducing anticonvulsants are eligible
14. Prior systemic anti-cancer (chemotherapy, immunotherapy, biologic therapy, vaccine) and investigational agents within 4 weeks or ≤ 5 x half-life of the agent (whichever is shorter) before first dose of capmatinib. If previous treatment is a monoclonal antibody, then the treatment must be discontinued at least 4 weeks before first dose of capmatinib. If previous treatment is an oral targeted agent, then the treatment must be discontinued at least 5 x half-life of the agent.
15. Impairment of GI function or GI disease that may significantly alter the absorption of capmatinib (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, or malabsorption syndrome)
16. Current or expected use of a prohibited medication as in Section 6.2.2 and Table 6-3.
17. Participants with known hypersensitivity to any of the excipients of capmatinib (crospovidone, mannitol, microcrystalline cellulose, povidone, sodium lauryl sulfate, magnesium stearate, colloidal silicon dioxide, and various coating premixes)
18. Any other condition that would, in the Investigator's judgment, contraindicate participant's participation in the clinical study due to safety concerns or compliance with clinical study procedures, e.g., active infection, inflammation, intestinal obstruction, unable to swallow medication, social/ psychological issues, etc.
19. Pregnant or nursing (lactating) women.
20. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and for 7 days after stopping treatment. Highly effective contraception methods include:

    * Total abstinence (when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
    * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) total hysterectomy, or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
    * Male sterilization (at least 6 months prior to screening). For female subjects on the study the vasectomized male partner should be the sole partner for that subject
    * Use of oral, injected or implanted hormonal methods of contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS), or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception. In case of use of oral contraception women should have been stable on the same pill for a minimum of 3 months before taking study treatment.

    Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g., age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks before study entry. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential
21. Sexually active males unless they use a condom during intercourse while taking drug and for 7 days after stopping treatment and should not father a child in this period. A condom is required for all sexually active male to prevent them from fathering a child AND to prevent delivery of study treatment via seminal fluid to partner. In addition, male participants must not donate sperm for the time period specified above
22. Patients who received live vaccines (e.g., intranasal influenza, measles, mumps, rubella, oral polio, BCG, yellow fever, varicella, TY21a typhoid vaccines and COVID 19 vaccines if a live COVID 19 vaccine becomes available) within 30 days prior to the first dose of IP.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-10-03 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
CNS Overall response rate (CORR) in | Up to 36 months
  Proportion of participants in with confirmed central nervous system complete response (CR) and/or partial response (PR) per RANO-BM criteria. CR: complete disappearance of all enhancing measurable and non-measurable disease sustained for at least 4 weeks; no new lesions; and stable or improved non-enhancing (T2/FLAIR) lesions. PR: ≥50% decrease, compared with baseline; the sum of products of perpendicular diameters of all measurable enhancing lesions sustained for at least 4 weeks; no progression of non-measurable disease; no new lesions; stable or improved non-enhancing (T2/FLAIR) lesions on the same or a lower dose of corticosteroids compared with baseline scan; and the patient being on a corticosteroid dose not greater than the dose at time of the baseline scan and stable or improved clinically.

SECONDARY OUTCOMES:
CNS Duration of response (DOR) | Up to 36 months
  Median time (months) from central nervous system (CNS) complete response (CR) or partial response (PR) until progressed disease (PD: ≥25% increase in lesion of perpendicular diameter), per RANO-BM criteria. CR: complete disappearance of all enhancing measurable and non-measurable disease sustained for at least 4 weeks; no new lesions; and stable or improved non-enhancing (T2/FLAIR) lesions. PR: ≥50% decrease, compared with baseline; the sum of products of perpendicular diameters of all measurable enhancing lesions sustained for at least 4 weeks; no progression of non-measurable disease; no new lesions; stable or improved non-enhancing (T2/FLAIR) lesions on the same or a lower dose of corticosteroids compared with baseline scan; and the patient being on a corticosteroid dose not greater than the dose at time of the baseline scan and stable or improved clinically.
CNS Progression-free survival (PFS) | Up to 36 months
  Median time (months) from central nervous system central nervous system complete response (CR) and/or partial response (PR) until progressive disease (PD) or death for the subjects whose best overall response CR or PR, per RANO-BM criteria. CR: complete disappearance of all enhancing measurable and non-measurable disease sustained for at least 4 weeks; no new lesions; and stable or improved non-enhancing (T2/FLAIR) lesions. PR: ≥50% decrease, compared with baseline; the sum of products of perpendicular diameters of all measurable enhancing lesions sustained for at least 4 weeks; no progression of non-measurable disease; no new lesions; stable or improved non-enhancing (T2/FLAIR) lesions on the same or a lower dose of corticosteroids compared with baseline scan; and the patient being on a corticosteroid dose not greater than the dose at time of the baseline scan and stable or improved clinically. PD: ≥25% increase in perpendicular diameter of any lesion.
CNS Overall response rate (CORR) (in cfDNA MET ex14 positive) | Up to 36 months
  Proportion of participants in with confirmed central nervous system complete response (CR) and/or partial response (PR) per RANO-BM criteria. CR: complete disappearance of all enhancing measurable and non-measurable disease sustained for at least 4 weeks; no new lesions; and stable or improved non-enhancing (T2/FLAIR) lesions. PR: ≥50% decrease, compared with baseline; the sum of products of perpendicular diameters of all measurable enhancing lesions sustained for at least 4 weeks; no progression of non-measurable disease; no new lesions; stable or improved non-enhancing (T2/FLAIR) lesions on the same or a lower dose of corticosteroids compared with baseline scan; and the patient being on a corticosteroid dose not greater than the dose at time of the baseline scan and stable or improved clinically.
Systemic Duration of Response (DOR) | Up to 36 months
  Median time (months) from systemic complete response (CR) or partial response (PR) until progressed disease (PD - ≥20% increase in sum of lesions), per RECISIT 1.1. Evaluation of Target Lesions (CR): the disappearance of all target lesions; any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR is at least a 30% decrease in the sum of the longest diameters of target lesions, taking as reference the baseline sum of the longest diameters. Evaluation of Non-target Lesions (CR): the disappearance of all non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological in size (<10 mm short axis). Non-CR / Non-PD: persistence of one or more non-target lesion(s) and/or the maintenance of tumor marker level above the normal limits.
Systemic Progression-free Surivial (PFS) | Up to 36 months
  Median time (months) from central nervous system central nervous system complete response (CR) and/or partial response (PR) until progressive disease (PD: ≥20% increase in sum of lesions) or death for the subjects whose best overall response CR or PR, per RECISIT 1.1. Evaluation of Target Lesions (CR): the disappearance of all target lesions; any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR is at least a 30% decrease in the sum of the longest diameters of target lesions, taking as reference the baseline sum of the longest diameters. Evaluation of Non-target Lesions (CR): the disappearance of all non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological in size (<10 mm short axis). Non-CR / Non-PD: persistence of one or more non-target lesion(s) and/or the maintenance of tumor marker level above the normal limits.
Systemic Objective response rate (ORR) | Up to 36 months
  Proportion of participants in with confirmed systemic complete response (CR) and/or partial response (PR) per RECISIT v1.1 criteria. Evaluation of Target Lesions (CR): the disappearance of all target lesions; any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR is at least a 30% decrease in the sum of the longest diameters of target lesions, taking as reference the baseline sum of the longest diameters. Evaluation of Non-target Lesions (CR): the disappearance of all non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological in size (<10 mm short axis). Non-CR / Non-PD: persistence of one or more non-target lesion(s) and/or the maintenance of tumor marker level above the normal limits.
Overall Survival (OS) | Up to 5 years
  Median time from either the date start of treatment that patients are still alive.
Overall response rate (ORR) | Up to 36 months
  The proportion of participants in with a confirmed complete response (CR) and/or partial response (PR) based on cross sectional imaging per RECIST 1.1. Evaluation of Target Lesions (CR): the disappearance of all target lesions; any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR is at least a 30% decrease in the sum of the longest diameters of target lesions, taking as reference the baseline sum of the longest diameters. Evaluation of Non-target Lesions (CR): the disappearance of all non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological in size (<10 mm short axis). Non-CR / Non-PD: persistence of one or more non-target lesion(s) and/or the maintenance of tumor marker level above the normal limits
Adverse Events (AEs) | Up to 36 months
  Incidence (frequency) of treatment-related adverse events (AEs) using NCI Common Terminology Criteria for Adverse Events (CTCAE, v.5.0)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy F Burns, MD, PhD, Principal Investigator — UPMC Hillman Cancer Center

IPD SHARING:
Plan to Share IPD: No